CLINICAL TRIAL: NCT05953818
Title: Changes of Cognitive Function and Brain Magnetic Resonance in Maintenance Hemodialysis Patients With Diabetes Mellitus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Collaborators: Beijing Shuyi Hospital (Other)
Responsible Party: Principal Investigator, Wenhu Liu, Clinical Professor, Beijing Friendship Hospital
Other Study IDs: 2022-P2-090-01
Record Dates: First submitted 2023-07-02; First posted 2023-07-20 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Maintenance Hemodialysis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Maintenance hemodialysis with diabetes group: The patients were given a quiet environment and completed the test within 10 minutes. The cognitive function of the two groups of patients was evaluated and analyzed using the Montreal Cognitive Assessment Scale (MoCA) in Chinese. The patients were given brain magnetic resonance high resolution structural imaging to observe changes in brain structure.
  Interventions: Diagnostic Test: Chinese version of the Montreal Cognitive Assessment Scale (MoCA) and brain magnetic resonance high resolution structural imaging
- Maintenance hemodialysis non diabetic group: The patients were given a quiet environment and completed the test within 10 minutes. The cognitive function of the two groups of patients was evaluated and analyzed using the Montreal Cognitive Assessment Scale (MoCA) in Chinese. The patients were given brain magnetic resonance high resolution structural imaging to observe changes in brain structure.
  Interventions: Diagnostic Test: Chinese version of the Montreal Cognitive Assessment Scale (MoCA) and brain magnetic resonance high resolution structural imaging

INTERVENTIONS:
Diagnostic Test: Chinese version of the Montreal Cognitive Assessment Scale (MoCA) and brain magnetic resonance high resolution structural imaging — Chinese version of Montreal cognitive assessment scale and brain magnetic resonance high resolution structural imaging

SUMMARY:
In recent years, due to the frequent occurrence of kidney disease and diabetes, the number of patients entering maintenance hemodialysis is increasing. With the economic development and dialysis quality improving year by year, the survival time of uremic patients is significantly prolonged, and the hazards of various complications are increasingly prominent. Cognitive impairment is a common complication of maintenance hemodialysis patients, and its specific mechanism is not yet clear. Type 2 diabetes mellitus (T2DM) and chronic kidney disease (CKD) are independent risk factors for cognitive impairment. The prevalence of cognitive impairment is higher in patients with type 2 diabetes and advanced chronic kidney disease, especially in patients with diabetes and end-stage renal disease (ESKD). T2DM and ESKD independently increase the risk of cerebrovascular disease and cognitive impairment. However, the relationship between diabetes mellitus and cognitive function in maintenance hemodialysis patients is unclear. However, compared with the general population, patients with type 2 diabetes mellitus (T2DM) and patients with advanced chronic kidney disease (CKD) had more severe brain atrophy, and the severity of white matter lesions on brain MRI increased. To sum up, the study of cognitive dysfunction is very important in maintenance hemodialysis patients with diabetes. It is urgent for us to explore the changes of cognitive impairment and brain magnetic resonance in maintenance hemodialysis patients with diabetes, so as to help detect brain cell damage and improve the survival rate and quality of life in the early stage of the disease.

DETAILED DESCRIPTION:
In recent years, due to the frequent occurrence of kidney diseases and diabetes, the number of patients entering maintenance hemodialysis is increasing. With the economic development and the improvement of dialysis quality year by year, the survival period of uremia patients is significantly prolonged, and the hazards of various complications are increasingly prominent. Cognitive dysfunction is a common complication of maintenance hemodialysis patients, and its specific mechanism is still unclear.

Firstly, let's talk about cognitive impairment and changes in brain magnetic resonance imaging.Cognitive function refers to the ability of the brain to perform advanced activities, including sensory perception, attention, memory, language, thinking, consciousness, and even emotions. Cognitive dysfunction is one or more aspects of the cognitive process that are impaired, mainly due to developmental and learning delays, brain trauma or brain diseases (such as stroke, brain trauma, Parkinson's disease, Alzheimer's disease, multiple sclerosis, schizophrenia, and other chronic diseases), or sociocultural conditions (such as malnutrition or environmental deprivation). Cognition is an important aspect of functional status and a determinant of patients' ability to control disease, live independently, and participate in nursing decision-making. Scholars have pointed out that patients' cognitive impairment is directly related to the degree of white matter injury, and is in direct proportion . Moreover, cognitive impairment can lead to changes in the hippocampus, gray matter, and white matter of the brain. Therefore, effective monitoring of the patient's brain, especially the white matter, is the key to implementing treatment. Brain magnetic resonance imaging can fully display the heterogeneity of water molecular dispersion in brain tissue. The new non-invasive three-dimensional arterial spin labeling (ASL) imaging technology provides a means to detect local hemodynamic changes. Compared to PET, its advantages lie in its non-invasive nature and rapid acquisition time under high magnetic field intensity (3.0 T).It can more effectively observe patients' early brain injury and diagnose early cognitive impairment. Previous studies have shown that for patients with early cognitive impairment, compared with healthy controls, MRI shows a symmetrical decrease in CBF values, mainly in the frontoparietal temporal lobe region, followed by marginal brain regions such as the cingulate gyrus and hippocampus, with the occipital lobe least affected.

Next, let's talk about cognitive impairment and changes in brain magnetic resonance imaging in maintenance hemodialysis patients. As a special group of people, maintenance hemodialysis (MHD) has been found to have widespread cognitive impairment. Tang Xiaojun's research found that the incidence of cognitive dysfunction in MHD patients can reach 61.84%, further proving that cognitive dysfunction is common in MHD populations. Once complicated with cognitive dysfunction, it not only seriously affects the treatment, daily life, and work of maintenance hemodialysis patients, but also affects their psychological status, nutritional status, and immune function, which may lead to poor prognosis such as death.

Cognitive dysfunction is affected by many aspects. Maintenance hemodialysis patients have many known risk factors for cognitive dysfunction, including risk factors associated with a variety of cardiovascular and cerebrovascular diseases and cardiovascular and cerebrovascular diseases, such as hypertension, diabetes and dyslipidemia, the neurotoxicity of uremic toxins, massive fluid and osmotic changes during dialysis, fluctuating uremic toxin titers. As MHD has become the main life-sustaining treatment for patients with end-stage renal disease (ESRD), the low perfusion volume caused by long-term MHD treatment will cause acute cerebral ischemia, and the decrease in cerebral blood flow is significantly associated with a decrease in overall and executive function and progress in the burden of white matter disease. Some studies have pointed out that the presence of cognitive impairment is one of the high-risk factors for adverse outcomes such as hospitalization, exacerbation, and termination of dialysis in MHD patients, while patients with cognitive impairment have a higher risk of death than patients without cognitive impairment. Therefore, early assessment of cognitive function and intervention therapy for MHD patients is of great significance. Because early symptoms of cognitive dysfunction are not obvious and it is difficult to attract attention from patients, it is necessary to observe the brain damage of patients as early as possible through magnetic resonance imaging methods to detect early cognitive dysfunction. Previous studies have shown that patients with ESRD undergo magnetic resonance imaging of the brain, and compared to normal individuals, the results suggest an increase in local cerebral blood flow (CBF), widespread gray matter atrophy, and a decrease in the volume of white matter in local brain regions. Moreover, maintenance hemodialysis may exacerbate brain atrophy in patients with ESRD, which is also accompanied by a decline in cognitive function.

Then let's talk about the cognitive dysfunction and brain MRI changes of diabetes patients. In recent years, with the rapid increase in the prevalence of diabetes and chronic kidney disease, the proportion of diabetes patients in hemodialysis patients in China is increasing. At present, a considerable number of diabetes patients have cognitive dysfunction, and in the coming decades, the number of diabetes patients with cognitive dysfunction will continue to increase. However, the hyperglycemia caused by diabetes will lead to increased plasma osmotic pressure, increased blood viscosity, and decreased metabolic rate of brain tissue, which will eventually lead to the reduction of local cerebral blood flow. In addition, diabetes patients have changes in microvascular basement membrane, extensive decline in neuronal function, and decline in brain metabolism, which can affect cognitive function. In 1966, Reske Nielsen carried out autopsy on 16 diabetes patients with cognitive impairment, and found that their brain tissue had severe diffuse degeneration of gray matter and white matter, and put forward the concept of "diabetes encephalopathy" for the first time.

Some studies believe that there is a relationship between cerebral perfusion and cognitive function in diabetes patients. Dai found that compared with the control group, diabetes patients had decreased cerebral blood flow in the resting default network, visual and cerebellar networks. The decline of blood flow in these brain regions was related to pleasure, memory, executive function, insulin resistance at baseline and cognitive dysfunction, indicating that diabetes patients had a correlation between resting local cerebral perfusion and cognitive function, and insulin resistance might promote the decline of local cerebral perfusion in diabetes patients.

Finally, let's talk about the cognitive dysfunction and brain MRI changes in patients with maintenance hemodialysis and diabetes. Type 2 diabetes (T2DM) and chronic kidney disease (CKD) are independent risk factors for cognitive dysfunction. The prevalence of cognitive dysfunction is higher in patients with type 2 diabetes and advanced chronic kidney disease, especially in patients with diabetes and end-stage kidney disease (ESKD). T2DM and ESKD independently increase the risk of cerebrovascular disease and cognitive impairment. The accumulation of advanced glycation end products in T2DM patients triggers vascular endothelial dysfunction, which may lead to more fragile and permeable cerebral blood vessels. However, the proinflammatory environment in ESKD patients causes vascular endothelial dysfunction and cerebral blood flow damage, leading to clinical and subclinical cerebrovascular diseases. Therefore, investigator speculate that T2DM may increase the risk of cognitive impairment in ESKD patients. However, there is currently limited data on the combined effects of T2DM and ESKD on neurocognition. Previous studies have shown that compared with patients without diabetes, MHD patients with diabetes have a significantly higher incidence of overall cognitive impairment, and perform poorly in overall cognition, visuospatial/executive function, naming, language, abstraction and orientation tasks. However, after adjusting multivariable factors, diabetes cannot independently predict the increased risk of overall cognitive impairment in MHD patients. Data on the relationship between diabetes and cognitive function in hemodialysis patients are still limited and controversial. The correlation between diabetes and cognitive function in MHD population is still unclear.

The situation of brain MRI in maintenance hemodialysis patients with diabetes is unknown at present. However, compared with the general population, brain atrophy is more serious in patients with type 2 diabetes (T2DM) and patients with advanced chronic kidney disease (CKD), and the severity of white matter lesions on brain magnetic resonance imaging (MRI) has increased.

To sum up, because cognitive dysfunction is related to the increased mortality of maintenance hemodialysis patients, compared with patients without cognitive dysfunction, patients with at least one cognitive impairment have a death risk of 77% or even higher, and type 2 diabetes may increase the risk of cognitive impairment in patients with end-stage renal disease. Therefore, the study of cognitive dysfunction in maintenance hemodialysis patients with diabetes is very important. It is urgent for investigator to explore the changes of cognitive dysfunction and brain magnetic resonance in maintenance hemodialysis patients with diabetes, so as to help detect brain cell damage at the early stage of disease and timely treatment, and improve the survival rate and quality of life of patients. Therefore, the purpose of this study was to analyze the changes of cognitive function and brain MRI in maintenance hemodialysis patients with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Age must be greater than 18 years old
* Receiving primary or higher education
* Dialysis 3 times a week, 4 hours per session, with dialysis time greater than 3 months
* Voluntarily participate in this study and sign an informed consent form.

Exclusion Criteria:Participants who meet any of the following conditions are excluded:

* The patient has any known Nervous system disease, such as dementia or Parkinson's disease.
* Have a history of mental illness, such as depression or schizophrenia.
* Suffering from visual, hearing, and language impairments, unable to cooperate with cognitive function assessment
* In the past 3 months, he has been unconscious, unconscious or other stress states due to infection, acute cardio cerebral Vascular disease.
* Suffering from severe liver damage or other serious physical diseases that may affect cognitive function.
* Have Alcohol dependence or psychotropic substance abuse, and currently use drugs that affect cognitive function or renal function.
* Patients with metallic substances in their bodies cannot pass magnetic resonance imaging (MRI) examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: During the period of 2023.01-2023.07 selection, 100 patients with complete and consistent data were collected from Beijing Friendship Hospital affiliated to Capital Medical University, Beijing Shunyi District hospital, and regular hemodialysis patients. According to whether they were diagnosed as diabetes, they were diabetic group and non-diabetic group respectively.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-05-30 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Brain magnetic resonance high-resolution structural imaging was performed to observe the changes of brain structure | 15 to 20 minutes
  All participants were examined with 3.0T MRI scanner (GE Healthcare, discovery mr750w, Milwaukee, WI), using quantitative techniques such as high-resolution structural magnetic resonance, resting state functional magnetic resonance and arteriovenous spin labeling imaging (ASL).

SECONDARY OUTCOMES:
The cognitive function of the two groups was evaluated and analyzed by the Chinese version of Montreal Cognitive Assessment Scale (MoCA) | 10 minutes
  The two groups of patients were given a quiet environment and completed the test within 10 minutes. The cognitive function of the two groups was evaluated and analyzed by the Chinese version of Montreal Cognitive Assessment Scale (MoCA). The possible score was between 0 and 30. The higher the score, the better the cognitive state. We defined cognitive impairment as a total score of less than 26 for participants with high school education or below and less than 27 for participants with high school education or above, because the average score of MOCA varies according to the level of education

CONTACTS AND LOCATIONS:
Overall Officials: Jia Wang, Principal Investigator — student
Locations (2):
- China (2):
  - Beijing Friendship hospital, Beijing, Beijing Municipality
  - Ethics Committee of Beijing Shunyi District Hosipital., Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No